CLINICAL TRIAL: NCT04522037
Title: Retrospective Study of the Measurement of the Efficacy of MORPHINE in the Early Management of Dyspnea in COVID-19 Positive Patients With Moderate to Severe Impairment Without Objective of Resuscitation Management (Level of Care 3 and 4) at the Hospices Civils of Lyon
Brief Title: Measurement of the Efficacy of MORPHINE in the Early Management of Dyspnea in COVID-19 Positive Patients
Acronym: CODYS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CODYS_2020
Record Dates: First submitted 2020-07-06; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-07

CONDITIONS: Patients Hospitalized in the Hospices Civils of Lyon; COVID-19 Disease; Moderate to Severe Dyspnea; Without Resuscitation Objective Management
Keywords: COVID-19 disease; level of care 3 and 4; morphinic treatment; dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interventional group: patients hospitalized at the hospices civils of Lyon with a level of care 3 or 4 receiving morphinic treatment for COVID-19 disease dyspnea.
  Interventions: Other: No intervention / Compare the difference in respiratory rate between H0 and H12 of the initiation of morphine between the control and interventional groups
- control group: patients hospitalized at the hospices civils of Lyon with a level of care 3 or 4 not receiving morphinic treatment for COVID-19 disease dyspnea.
  Interventions: Other: No intervention / Compare the difference in respiratory rate between H0 and H12 of the initiation of morphine between the control and interventional groups

INTERVENTIONS:
Other: No intervention / Compare the difference in respiratory rate between H0 and H12 of the initiation of morphine between the control and interventional groups — Respiratory rate is analyzed with the scope (approved by the French national medical authorities)

SUMMARY:
Morphine is used in the treatment of dyspnea and polypnea with a proven benefit on the improvement of these symptoms, both etiologically and symptomatically. This medication is used in particular in palliative care for this type of symptom.

The Sars CoV2 viral pneumonia table can lead to respiratory distress. In patients with moderate to severe impairment without goal of resuscitation (level of care 3 and 4), the introduction of morphine may sometimes be necessary to relieve respiratory symptoms. These also lead to major exhaustion which can worsen the clinical picture. However, the prescription of morphine is not systematic in front of a respiratory distress table.

The investigators hypothesized that early treatment with morphine lead to a better management of dyspnea, quality of live and survival in COVID-19 positive participants patients when there is not resuscitation objective management (level of care 3 and 4).

The objective is to measure the efficacy of morphine in the early management of dyspnea, quality of life and survival in COVID-19 positive participants patients treated in the Hospices Civils of Lyon during COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Having had a Covid-19 respiratory disease confirmed by PCR or TDM or anamnestic criterion for patients living in communities for the elderly (respiratory symptomatology suggestive and at least 3 cases confirmed in the living environment).
* Having had respiratory severity criteria: respiratory distress syndrome including FR> 25 / min and oxygen-demand> 4 L / min to maintain a SpO2> 90% at inclusion.
* Having had a defined level of care after collegial discussion notified in the file rejecting the external cardiac massage and admission to the intensive care unit (Level 3 and 4 on the protocols of the Hospices Civils de Lyon).
* Collection of non-opposition

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized at the hospices civils of Lyon with a level of care 3 or 4 receiving morphinic and not receiving morphinic treatment for COVID-19 disease dyspnea.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Title : Reduction of respiratory rate between Hour 0 and Hour 12 at initiation of morphine treatment | Hour 0 and Hour 12 after initiation of morphinic treatment
  The respiratory rate is analyzed at Hour 0 and Hour 12 by a scope.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital de la Croix Rousse / GHN, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Lyon Sud, Pierre-Bénite